CLINICAL TRIAL: NCT06314750
Title: Deep Learning Based MRI Radiomics in Predicting the Clinical Risk of Locally Advanced Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Cai Zerong, Deputy Director of the Department, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2023ZSLYEC-680
Record Dates: First submitted 2024-03-09; First posted 2024-03-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced Rectal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The pathological specimens before operation and the specimens after operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Well T-downstage: After receiving neoadjuvant therapy, the postoperative pathological stage of patients with primary cT4 rectal cancer was pT2 or less.
- Poor T-downstage: After receiving neoadjuvant therapy, the postoperative pathological stage of patients with primary cT4 rectal cancer was pT3 or above.

SUMMARY:
Neoadjuvant therapy is the standard diagnosis and treatment strategy for locally advanced rectal cancer defined by MRI in order to achieve tumor regression, thus affecting the selection of surgical strategy and circumferential margin, improving the safety of operation and the prognosis of patients. This study focused on the related clinical factors such as tumor regression before and after neoadjuvant therapy, combined with preoperative high-dimensional features such as radiomics, to predict the related factors of tumor regression of locally advanced rectal cancer, and validate it with multicenter. In order to develop an accurate model that can be applied to the real world and stratify the risk of locally advanced rectal cancer patients before treatment.

DETAILED DESCRIPTION:
The patients with locally advanced rectal cancer were collected retrospectively, and the relevant information such as clinical baseline characteristics, imaging data and preoperative/postoperative pathological data were collected and integrated, applying the method of deep learning to construct the model, in order to predict and evaluate the risk factors (invasion of mesorectal fascia, status of cancer nodule, long-term prognosis, tumor recurrence, etc.) which are important in clinical diagnosis and treatment. After the model was established, prospective studies were carried out to validate the model, continue training and enrich the effectiveness of the model.

ELIGIBILITY:
Inclusion Criteria:

1. Primary rectal adenocarcinoma was diagnosed before operation
2. Preoperative MRI staging was diagnosed as stage cT4 rectal cancer
3. Receiving neoadjuvant therapy before operation (including but not limited to chemotherapy, radiotherapy, immunotherapy or targeted therapy, etc.)
4. Middle and low rectal cancer (the distance between the lower margin of the tumor and the anal margin ≤ 12cm measured by MRI)
5. Receive radical resection of rectal cancer

Exclusion Criteria:

1. lack of clinical TNM staging information or other key clinical information about MRI
2. the imaging quality is poor or the MRI image has artifacts

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 136 patients (Well T-downstage: 28.68%, 39/136) were included in the training cohort and 50 (Well T-downstage: 30%, 15/50) patients in the test cohort.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 120 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Zerong Cai, MD, Study Director — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No
Please contact us by Email